CLINICAL TRIAL: NCT05227157
Title: Comparison of the Perception of Metallic Taste According to Lingual Locations in Healthy Volunteers
Brief Title: GOUTMETALSAIN: Comparison of the Perception of Metallic Taste According to Lingual Locations in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Valence (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH-CHV-10
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Taste Disorders; Sensation Disorders; Taste, Metallic; Taste Disorder, Glossopharyngeal Nerve
Keywords: Taste, Metallic
MeSH Terms: conditions — Taste Disorders; Sensation Disorders; Glossopharyngeal Nerve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: intensity of perception of metallic taste: For this study, there is only one arm: swab with iron sulfate solution at a concentration of 10g/l.
  Each subject complete visual scale
  Interventions: Other: swab with iron sulfate solution

INTERVENTIONS:
Other: swab with iron sulfate solution — measurement of the intensity of perception of metallic taste by affixing a swab iron sulfate solution 10g/l at 4 places on the tongue depending on the glossopharyngeal nerve: tip of the tongue (right and left); base of the tongue (right and left). Visual analogic Scale (0 to 5)

SUMMARY:
This is a mono center , observational study carried out within otorhinolaryngology department in CH Valence.

This is a descriptive and exploratory study in healthy volunteers. Based on the hypothesis that Metallic taste is imperfectly assessed, this study will provide a better understanding of the Metallic Taste.

DETAILED DESCRIPTION:
The study consists of the application of a swab soaked in iron sulfate at a concentration of 10g/l.

each patient will rate the intensity he/she perceives (on a numerical scale from 1 to 5) at each of the 4 predefined lingual locations

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Healthy volunteers
* Read, write and understand the French language
* Patient affiliated to a social security system
* Written and signed informed consent

Exclusion Criteria:

* head and Neck cancer history
* olfactory and gustatory disorder
* Refusal to participate in research
* Patient under guardianship, deprived of liberty, safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volonteers without olfactory and gustatory disorder
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
evaluation of the intensity of metallic taste | 5 minutes
  visual analogue scale (0 to 5); A score of 5 means the highest intensity of metallic taste

CONTACTS AND LOCATIONS:
Locations (1):
- Ch Valence, Valence, Drome, France